CLINICAL TRIAL: NCT05338424
Title: Sprint Interval Training to Target Brain Oscillations in Psychosis
Brief Title: Exercise Target Brain Oscillations in Psychosis
Status: Withdrawn | Type: Observational
Why Stopped: Principal Investigator left the institution
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: PSYCH-2022-30666
Record Dates: First submitted 2022-04-04; First posted 2022-04-21 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Psychosis; Schizophrenia; Schizoaffective Disorder
Keywords: Psychosis; Schizophrenia; Schizoaffective Disorder; Exercise; Cognition; Attention
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sprint Interval Training (SIT): The 1-session SIT protocol will include "Work" bouts performed at maximal intensity targets. Three "Work" bouts will be performed at 20-second intervals separated by 2 recovery bouts consisting of 2 minutes of low-intensity cycling. The SIT session will employ a standardized warm up and cool down of 3 minutes at a self-selected light intensity, per current guidelines. SIT sessions will take 15 minutes to complete.
  Interventions: Other: Sprint Interval Training (SIT)
- Stretching: Stretching will include a low-intensity range of motion and stretching exercises with session duration (15 minutes) being matched to SIT.

INTERVENTIONS:
Other: Sprint Interval Training (SIT) — Active arm-- exercise dictated by protocol
  Groups: Sprint Interval Training (SIT)

SUMMARY:
Previous studies have shown that cardiorespiratory fitness (how well the heart and lungs are able to function during physical activity) is often reduced in people with psychosis. The goal of this research study is to test the hypothesis that aerobic exercise can lead to small changes in brain functioning that can influence visual perception and attention in psychosis. The type of aerobic exercise used in this study is called Sprint Interval Training, or "SIT". Information from this study will help to develop interventions that enhance cognition and maximize the quality of life for persons living with psychosis.

The exercise procedure used is called SIT, which involves training rigorously on a stationary bike for a short period of time followed by a resting period.

ELIGIBILITY:
Inclusion Criteria:

* Meet diagnostic criteria for schizophrenia or schizoaffective disorder
* Are age 18-64
* Fluent in written and spoken English
* Have an outpatient status of at least 1 month prior to participation
* Has been on a stable dose of psychiatric medication for at least one month prior to participation (titration to a lower dose of psychotropic medications under supervision of a psychiatrist can be allowed at the discretion of the investigators)

Exclusion Criteria:

* Current or possibility of current pregnancy (self-reported)
* Active suicidal ideation at screening or baseline assessments, or previous intent to act on suicidal ideation with a specific plan, preparatory acts, or an actual suicide attempt within the last 3 months, as indicated by the C-SSRS
* WTAR standardized score below 70
* American College of Sports Medicine contraindication to exercise

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Individuals in good health with a psychotic disorder.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Individual Alpha Frequency | through study completion, on average 2 weeks
  A prominent neural oscillatory rhythm measured from resting EEG.
Change in Visual Attention | through study completion, on average 2 weeks
  Computerized tasks that measure speeded sustained attention.
Change in Visual Perception | through study completion, on average 2 weeks
  Computerized tasks that measure speeded visual perception

CONTACTS AND LOCATIONS:
Overall Officials: Ian Ramsay, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States